CLINICAL TRIAL: NCT05223244
Title: Bladder Capacity as an Objective Measure of Response to Intravesical Treatment of Newly Diagnosed Interstitial Cystitis: a Prospective, Randomized Trial
Brief Title: Bladder Capacity as Objective Measure of Intravesical Treatment of Newly Diagnosed IC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Adam Gafni-Kane, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EH11-081
Record Dates: First submitted 2022-01-24; First posted 2022-02-03 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: dimethyl sulfoxide (DMSO); Intravesical instillations; bupivacaine, triamcinolone, and heparin (BTH); Bladder instillations
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Bupivacaine; Triamcinolone; Heparin; Dimethyl Sulfoxide

STUDY DESIGN:
Intervention Model Description: At each of the six weekly treatment visits, bladder capacity was determined, followed by the intravesical treatment of either DMSO or BTH.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients, investigators, and outcomes assessors were blinded to treatment patients received
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dimethyl sulfoxide (DMSO) (Active Comparator): Six weekly bladder instillations with 50mL of DMSO and 1mL of triamcinolone (10mg/mL)
  Interventions: Drug: dimethyl sulfoxide (DMSO)
- bupivacaine, triamcinolone, and heparin (BTH) (Experimental): Six weekly bladder instillations with 30mL of 0.5% bupivacaine (5mg/mL), 2mL triamcinolone (10mg/mL), and 2mL Heparin (10,000units/mL)
  Interventions: Drug: bupivacaine, triamcinolone, and heparin (BTH)

INTERVENTIONS:
Drug: bupivacaine, triamcinolone, and heparin (BTH) — 30mL of 0.5% bupivacaine (5mg/mL), 2mL triamcinolone (10mg/mL), and 2mL Heparin (10,000units/mL)
  Arms: bupivacaine, triamcinolone, and heparin (BTH)
Drug: dimethyl sulfoxide (DMSO) — 50mL of DMSO and 1mL of triamcinolone (10mg/mL)
  Arms: dimethyl sulfoxide (DMSO)

SUMMARY:
A comparative study of subjective outcomes following intravesical treatment of interstitial cystitis (IC) is lacking in the literature. Furthermore, an objective measure to determine the efficacy of intravesical treatment for interstitial cystitis has yet to be defined. Change in bladder capacity following therapy has been investigated; however, a formal statistical analysis of its utility in determining efficacy has yet to be performed. The primary objective of this prospective, randomized study is to determine whether there is a significant difference in subjective improvement in IC symptoms in women with newly diagnosed IC when treated with either dimethyl sulfoxide (DMSO) or bupivacaine, triamcinolone, and heparin (BTH) instillations. The secondary objective is to determine whether change in bladder capacity can be used as an objective measure of response to intravesical therapy for newly diagnosed interstitial cystitis. Our long-term goals are to improve the scientific understanding of therapy for interstitial cystitis, to improve patient counseling prior to initiation of treatment, and to better identify patients likely to receive inadequate relief of symptoms following intravesical treatment so that an alternative treatment can be pursued.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed interstitial cystitis/painful bladder syndrome

Exclusion Criteria:

* History of pelvic radiation, a history of bladder cancer, or a history of bladder resection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2011-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Reduction of at least 29.5% in ICSI score | 6 weeks
  reduction of at least 29.5% in ICSI score

SECONDARY OUTCOMES:
Bladder capacity | 6 weeks
  measurement of bladder capacity as determined by retro fill volume